CLINICAL TRIAL: NCT01594450
Title: Use of Biological Mesh Versus Standard Wound Care in Infected Incisional Ventral Hernias: a Multicenter Randomized Controlled Trial, the SIMBIOSE Study
Brief Title: Biological Meshes in Infected Fields: a Randomized Controlled Trial
Acronym: SIMBIOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011_56; 2011-A00059-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2012-04-22; First posted 2012-05-09 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2019-08

CONDITIONS: Ventral Hernia
Keywords: incisional ventral hernia; infected field; biological mesh
MeSH Terms: conditions — Hernia, Ventral | interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biological mesh (Experimental): patients will undergo the implantation of a biological mesh (after debridement and treatment of the infection) at the same time as the primary operation, or within one month of randomization.
  Interventions: Biological: Biological mesh
- without biological mesh (Active Comparator): patients undergo traditional wound care (debridement and treatment of infection), without placement of a biological mesh. For arm B, the common wound care used follows the normal practice of the treating surgeon, except the placement of the biological mesh, which must not be performed within 6 months of randomization.
  Interventions: Procedure: without biological mesh

INTERVENTIONS:
Biological: Biological mesh — patients will undergo the implantation of a biological mesh (after debridement and treatment of the infection) at the same time as the primary operation, or within one month of randomization.
  Other Names: Biologics; Acellular dermal matrix
  Arms: biological mesh
Procedure: without biological mesh — patients undergo traditional wound care (debridement and treatment of infection), without placement of a biological mesh. For arm B, the common wound care used follows the normal practice of the treating surgeon, except the placement of the biological mesh, which must not be performed within 6 months of randomization In cases of treatment failure at 6 months, patients of arm B are allowed to undergo any treatment which the treating surgeon views suitable, including a surgical procedure with implantation of a biological mesh
  Other Names: standard wound care
  Arms: without biological mesh

SUMMARY:
The SIMBIOSE trial is a large multicenter phase III prospective randomized controlled single blinded trial comparing the use of biological mesh versus traditional wound care without biological mesh in patients with an infected incisional ventral hernia. The primary endpoint is 6-month infectious and/or wound morbidity. Secondary endpoints are wound infection rate at 45 days, 3 months and 1 year, recurrent hernia rates at 1, 2 and 3 years, postoperative pain, quality of life, time to healing, need for wound reoperation, impact of the cross-linked mesh structure, and medico-economic evaluation. One hundred patients need to be included.

DETAILED DESCRIPTION:
Comparison between standard wound care and the use of biological meshes in infected fields

ELIGIBILITY:
Inclusion Criteria:

* wound infection related to a synthetic non-absorbable mesh for at least 15 days duration
* incisional abdominal hernia with an abcess or fistula, without the presence of a synthetic non-absorbable mesh
* incisional abdominal hernias smaller than 20 centimeter in the 2 largest diameters
* incisional abdominal hernias requiring a surgical procedure
* incisional abdominal hernias amenable to repair with a single biological mesh
* age over 18 years

Exclusion Criteria:

* non-infected incisional abdominal hernia
* history of biological mesh placement
* incisional abdominal hernia in contaminated, but non infected field (stoma presence, violation of gastrointestinal tract)
* incisional abdominal hernia larger than 20 x 20 cm
* BMI ≥ 40 kg/m2
* ASA score 4 and 5
* immunosuppression (including steroid and cytotoxic therapy)
* chronic disease such as cirrhosis, renal insufficiency with renal dialysis, malignant disease, known collagen disorder
* life expectancy under than 36 months
* allergy to one of the biological mesh components
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
6-month postoperative morbidity | 6 months

SECONDARY OUTCOMES:
Day 45 wound infection rate | 45 days
1-year recurrent hernia rates | 1 year
postoperative pain | up to 3 years
quality of life | up to 3 years
time to cure | up to 3 years
need for wound reoperation due to infection or hernia recurrence | up to 3 years
impact of the cross-linked mesh structure on the primary objective | 6 months
medico-economic evaluation taking into account direct costs related to infected ventral hernia treatment. | up to 3 years
3 months wound infection rate | 3 months
1 year wound infection rate | 1 year
2-year recurrent hernia rates | 2 years
3-year recurrent hernia rates | 3 years
impact of the cross-linked mesh structure on the 1-year infection rate | 1 year
impact of the cross-linked mesh structure on the 1-year recurrence rate | 1 year
impact of the cross-linked mesh structure on the 3-year recurrence rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Piessen, MD, PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Claude Huriez Hospital, University hospital, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mariette C, Briez N, Denies F, Dervaux B, Duhamel A, Guilbert M, Bruyere E, Robb WB, Piessen G; FRENCH. Use of biological mesh versus standard wound care in infected incisional ventral hernias, the SIMBIOSE study: a study protocol for a randomized multicenter controlled trial. Trials. 2013 May 7;14:131. doi: 10.1186/1745-6215-14-131. PMID 23782773